CLINICAL TRIAL: NCT01719835
Title: CHEMO-T: Cyclophosphamide, Doxorubicin, Vincristine and Prednisolone (CHOP) Versus Gemcitabine, Cisplatin and Methyl Prednisolone (GEM-P) in the First Line Treatment Of T-cell Lymphoma,a Multicentre Randomised Phase II Study
Brief Title: CHOP vs GEM-P in 1st Line Treatment of T-cell Lymphoma, Multicentre Phase II Study
Acronym: CHEMO-T
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMH CCR: 3549; 2011-004146-18 (EudraCT Number)
Record Dates: First submitted 2012-04-12; First posted 2012-11-01 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Peripheral T-cell Lymphoma NOS; Anaplastic Large Cell Lymphoma, ALK-Negative; Angioimmunoblastic T-cell Lymphoma; Hepatosplenic Gamma/ Delta T-cell Lymphoma; Enteropathy-Associated T-Cell Lymphoma
Keywords: T-Cell Lymphoma; Untreated
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Enteropathy-Associated T-Cell Lymphoma | interventions — Cyclophosphamide; Gemcitabine; Doxorubicin; Vincristine; Prednisolone; Methylprednisolone; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy GEM-P (Experimental): Gemcitabine, Methylprednisolone, Cisplatin
  Interventions: Drug: Gemcitabine; Drug: methylprednisolone; Drug: Cisplatin
- Chemotherapy CHOP (Active Comparator): Cyclophosphamide, Doxorubicin, Vincristine, Prednisolone
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone

INTERVENTIONS:
Drug: Cyclophosphamide — 750mg/m2 IV every 21 days
  Arms: Chemotherapy CHOP
Drug: Gemcitabine — 1000mg/m2 IV Days 1, 8, 15 every 28 days
  Arms: Chemotherapy GEM-P
Drug: Doxorubicin — 50mg/m2 IV every 21 days
  Arms: Chemotherapy CHOP
Drug: Vincristine — 1.4mg/m2 (max 2mg) IV every 21 days
  Arms: Chemotherapy CHOP
Drug: Prednisolone — 100mg PO Days 1-5 every 21 days
  Arms: Chemotherapy CHOP
Drug: methylprednisolone — 1000mg oral or IV Days 1-5 every 28 days
  Arms: Chemotherapy GEM-P
Drug: Cisplatin — 100mg/m2 IV Day 15 every 28 days
  Arms: Chemotherapy GEM-P

SUMMARY:
This is a randomised, open-label phase II study comparing GEM-P chemotherapy (experimental arm) with CHOP (control arm) in previously untreated T-cell lymphoma. Eligible patients will be randomised 1:1 between 4-weekly GEM-P or 3-weekly CHOP chemotherapy.

DETAILED DESCRIPTION:
Background:

T-cell lymphoma is an aggressive rare subset of Non-Hodgkin lymphoma (NHL) comprising several different subtypes of disease within this group. No standard first-line treatment exists for T-cell lymphoma as published series are small, with heterogeneous populations and often retrospective.

Protocol Synopsis, Study Period: 5 years

Objectives:

Primary:

• To compare the complete response rate of GEM-P with CHOP chemotherapy in the first line treatment of patients with T-Cell Lymphoma.

Secondary:

To investigate, between both arms:

* Rate of metabolic complete response
* Toxicity of treatment
* Overall survival (OS)
* Progression Free Survival (PFS)

Exploratory:

• Investigate impact of International Prognostic Index (IPI) on the outcomes response rate, PFS and OS

Study Design:

A randomised multi-centre open-label phase II study

Indication: Previously untreated T-Cell lymphoma No of Participants: 186 (93 patients in each arm)

Main Eligibility Criteria:

* Histologically proven T-cell lymphoma of the following subtypes:
* Peripheral T-cell lymphoma NOS
* Systemic Anaplastic large cell lymphoma (ALCL) Anaplastic lymphoma kinase (ALK) negative cases only
* Angioimmunoblastic T-cell lymphoma
* Hepatosplenic gamma/ delta T-cell lymphoma
* Enteropathy-associated T-cell lymphoma
* Bulky Stage I, Stage II, III or IV
* No prior chemotherapy regimen
* Patients aged 18 years or over.
* WHO performance status 0,1 or 2
* Adequate organ function:
* No Central Nervous System(CNS) or leptomeningeal involvement with lymphoma
* No treatment for lymphoma within 4 weeks of commencing trial therapy
* No known HIV, active Hepatitis B or C infection

Treatment:

CHOP: cyclophosphamide, doxorubicin, vincristine, prednisolone every 21 days. GEM-P: gemcitabine, methylprednisolone, cisplatin every 28 days.

Assessment Schedule:

* Patients will be reviewed at baseline and prior to each scheduled dose of treatment for toxicity
* Radiological tumour assessment will be done with CT scan after every 2 cycles in Arm A and after cycle 1, 3 and 4 in Arm B
* PET/CT scan will be performed at baseline and upon completion of treatment..
* Follow up after completion of treatment will be 3, 6, 9, 12, 18, 24 months then annually for 5 years in total. CT scan will be performed at 3 & 12 months.
* Following disease progression patients will be followed for survival every 3 months until death

ELIGIBILITY:
Inclusion Criteria:

Previously untreated, histologically proven T-cell Lymphoma (any of the following):

* Peripheral T-cell lymphoma Not Otherwise Specified (PTCL NOS)
* Systemic Anaplastic large cell lymphoma (ALCL) ALK negative cases only
* Angioimmunoblastic T-cell lymphoma
* Hepatosplenic gamma/ delta T-cell lymphoma
* Enteropathy-associated T-cell lymphoma (EATL)

  * Bulky stage I not being considered for reduced chemotherapy plus involved field radiotherapy or stage II, III or IV.
  * Patient is male or female, and ≥18 years of age on the day of signing informed consent.
  * WHO performance status 0, 1 or 2.
  * Cross sectional imaging from a baseline contrast enhanced CT should show at least one measurable disease site that is at least 2 cm in longest diameter and measurable in two perpendicular dimensions with or without corresponding Fluorodeoxyglucose(FDG) avid lesions.
  * Adequate cardiac function; formal assessment of left ventricular ejection fraction is only required if clinically indicated (a baseline echocardiogram should be done for patients with either hypertension, age > 60 years or history of cardiac disease)
  * Adequate bone marrow function: absolute neutrophil count (ANC) ≥1.0x109/l; white blood cell count ≥ 3x109/l; platelets ≥ 100x109/l; haemoglobin (Hb) ≥ 9g/dl (can be post-transfusion), unless deemed disease related
  * Adequate renal function: calculated creatinine clearance ≥50ml/minute.
  * Adequate liver function: serum bilirubin ≤1.5x Upper limit of normal (ULN); Alanine transaminase/Aspartate transaminase (ALT/AST) ≤2.5x ULN; ALP ≤3x ULN (in the absence of liver metastases). If liver metastases are present, ALT, AST or Alkaline phosphatase (ALP) ≤5x ULN are permitted. Isolated hyperbilirubinaemia due to Gilbert's disease is acceptable
  * Female patient of childbearing potential must have a negative serum or urine β-human chorionic gonadotropin(hCG)pregnancy test at baseline.
  * Written informed consent must be obtained prior to start of study treatments. Scans and bone marrow biopsies performed within 4 weeks of commencement of therapy will be acceptable provided they have been performed according to study requirements.
  * Patient agreeable to use contraception for the period of study treatment and up to 12 months after the last dose of study drugs.

Exclusion Criteria:

* Documented or symptomatic central nervous system involvement or leptomeningeal disease.
* Patients with no measurable disease on the contrast enhanced CT scan at baseline.
* Any other clinically significant disease or co-morbidity which may adversely affect the safe delivery of treatment within this trial.
* Any other malignancies diagnosed or treated within the last 5 years (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix).
* Treatment with another investigational agent within 30 days of commencing study treatment.
* Known positive tests for human immunodeficiency virus (HIV) infection, hepatitis C virus, acute or active hepatitis B infection.
* Patient is pregnant or breastfeeding, or expecting to conceive or father children within one year of finishing study treatment.
* Patients with poorly controlled diabetes mellitus
* Hypersensitivity or contraindication to any of the study drugs as stated in the Summaries of product characteristics(SmPCs)for each of the study drugs. Patients with previous cardiac infarct but satisfactory cardiac function may be allowed at the discretion of Chief Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-03; Primary Completion 2016-11-30 (Actual); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
complete response rate (CR/CRu) | approximately 20 weeks after randomisation

SECONDARY OUTCOMES:
Toxicity | approximately 20 weeks after randomisation
  using Common Terminology Criteria for Adverse Events (CTCAE)v4.0
Overall Survival | 1 and 2 years
Progression Free survival | 1 and 2 years
Metabolic Complete Response Rate | approximately 20 weeks after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, MD FRCP, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust - London and Surrey, London, United Kingdom

REFERENCES:
- [Derived] Gleeson M, Peckitt C, To YM, Edwards L, Oates J, Wotherspoon A, Attygalle AD, Zerizer I, Sharma B, Chua S, Begum R, Chau I, Johnson P, Ardeshna KM, Hawkes EA, Macheta MP, Collins GP, Radford J, Forbes A, Hart A, Montoto S, McKay P, Benstead K, Morley N, Kalakonda N, Hasan Y, Turner D, Cunningham D. CHOP versus GEM-P in previously untreated patients with peripheral T-cell lymphoma (CHEMO-T): a phase 2, multicentre, randomised, open-label trial. Lancet Haematol. 2018 May;5(5):e190-e200. doi: 10.1016/S2352-3026(18)30039-5. PMID 29703335